CLINICAL TRIAL: NCT01908153
Title: Taste Reward Processing in Pediatric Obesity
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cara Bohon, PhD, Assistant Professor, Stanford University
Other Study IDs: UL1TR000093 (NIH)
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Pediatric Obesity
Keywords: Picture food type; Taste type
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Overweight/Obese: Children with BMI percentile of 85 or above.
- Healthy Weight: Children with BMI percentile between 15 and 85.

SUMMARY:
The study aims to provide a better understanding of the neural influence of eating behavior in the development of childhood obesity. Children ages 4-8 will be recruited to examine fMRI brain response to pictures that signal delivery of a chocolate milkshake and to the taste itself. The brain response will be compared to body mass index percentile scores for each child to help us determine whether brain differences present in adolescents and adults with obesity are present in young children.

ELIGIBILITY:
Inclusion Criteria:

* ages 4-8
* parent available to complete surveys in English

Exclusion Criteria:

* no presence of metal in body
* no claustrophobia
* no psychiatric or neurological condition that will affect brain function

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 4-8
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
fMRI brain response to taste of chocolate milkshake | Baseline
fMRI brain response to picture cue | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cara Bohon, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Department of Psychiatry, Stanford, California, United States

REFERENCES:
- [Result] Bohon C. Brain response to taste in overweight children: A pilot feasibility study. PLoS One. 2017 Feb 24;12(2):e0172604. doi: 10.1371/journal.pone.0172604. eCollection 2017. PMID 28235080